CLINICAL TRIAL: NCT05858645
Title: Correction of Psoriatic T Cell Signatures by Deucravacitinib
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-37660
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- deucravacitinib treatment (Experimental): treatment with deucravacitinib for 6 months
  Interventions: Drug: deucravacitinib

INTERVENTIONS:
Drug: deucravacitinib — Treatment with deucravacitinib, skin biopsy and blood analysis pre- and mid-treatment

SUMMARY:
This study aims to assess cutaneous and blood immune cell function of patients with psoriasis before and after initiation of treatment with the Tyrosine kinase 2 (TYK2) blocker, deucravacitinib.

DETAILED DESCRIPTION:
This is a one-arm, open-label study to examine the effect of deucravacitinib on cutaneous and blood immune cells of psoriatic patients. 25 subjects with moderate to severe psoriasis will be enrolled. Biopsy and blood samples will be collected before and during treatment and undergo molecular profiling to assess for deucravacitinib-corrected signatures.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Patients with moderate-severe psoriasis (BSA >= 10%, PASI >=12, static Physician's Global Assessment (sPGA) 3 and above)

Exclusion Criteria:

1. taking systemic immunosuppressives in the last 12 weeks
2. pregnancy
3. severe immunodeficiency (either from genetic or infectious causes).
4. tuberculosis or other active serious infection
5. active systemic malignancy.
6. breast-feeding
7. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Psoriasis Area and Severity Index (PASI) score | pre-treatment, 4 months
  Change in severity and extent of psoriasis (calculated by Psoriasis Area and Severity Index (PASI) score); scale range of 0 to 72, 72 being maximal disease

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Cho, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No